CLINICAL TRIAL: NCT00650572
Title: A Study of ARRY-380 in Patients With Advanced HER2+ Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-380-101
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Cancer
Keywords: human epidermal growth factor receptor 2; epidermal growth factor receptor; EGFR; type I receptor tyrosine kinase
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARRY-380 (Experimental)
  Interventions: Drug: ARRY-380, HER2 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-380, HER2 inhibitor; oral — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule.

SUMMARY:
This is a Phase 1 study during which patients with advanced HER2+ solid malignancies or HER2+ metastatic breast cancer will receive investigational study drug ARRY-380.

This study has 2 parts. In the first part, patients with advanced HER2+ solid malignancies, who have already received at least one previous standard therapy, will receive increasing doses of study drug in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Approximately 30 patients from the US will be enrolled in Part 1 (Completed).

In the second part of this study, patients with HER2+ metastatic breast cancer, who have already received at least one previous standard therapy, will receive the best dose of study drug determined from the first part of the study and will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 20 patients from the US will be enrolled in Part 2 (Active, not recruiting).

ELIGIBILITY:
Key Inclusion Criteria (Part 1 and Part 2):

* Histological or cytological evidence of HER2+ cancer (Part 1) or HER2+ metastatic breast cancer (Part 2).
* Patients should have received at least one previous therapeutic regimen and either no longer are candidates for standard therapy, have no standard therapy available, or choose not to pursue standard therapy (patients with HER2+ breast cancer and with clinical indication for trastuzumab or lapatinib should have received prior therapy with trastuzumab and lapatinib, if available).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) between 0 and 2.
* Additional criteria exist.

Key Exclusion Criteria (Part 1 and Part 2):

* Uncontrolled or symptomatic brain metastases (patients may be considered adequately controlled if on a stable steroid dose for at least 30 days).
* Treatment with an investigational medicinal product or device within 30 days prior to first dose of study drug.
* Radiotherapy within 28 days prior to first dose of study drug (not including palliative radiotherapy at focal sites).
* Chemotherapy within 21 days prior to first dose of study drug.
* Major surgery within 30 days prior to first dose of study drug.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or active hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1, one year; Part 2, one year
Establish the maximum tolerated dose (MTD) of the study drug. | Part 1, one year
Characterize the pharmacokinetics of the study drug. | Part 2, one year
Assess amplification/expression of HER2 in archival and tumor tissues. | Part 2, one year

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of the study drug. | Part 1, one year
Assess changes in tumor markers. | Part 1, one year
Assess the efficacy of study drug in terms of tumor response and duration of response. | Part 1, one year; Part 2, one year
Assess expression of growth factor pathway proteins in archival and tumor tissues. | Part 2, one year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - The University of Colorado Cancer Center, Aurora, Colorado
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario